CLINICAL TRIAL: NCT00835835
Title: Lokomat Treadmill Training Effects on MS Gait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Jennifer Ruiz, DPT, Research Manager, Mount Sinai Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AL0001
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Gait, Unsteady; Multiple Sclerosis
Keywords: Multiple Sclerosis; gait; falls; lokomat; body-weight support treadmill training
MeSH Terms: conditions — Gait Disorders, Neurologic; Multiple Sclerosis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Placebo Comparator): The placebo group did not receive treatment during the matched period yet did undergo all assessments. The MS Placebo group received equal treatment following the study intervention period.
  Interventions: Other: Usual Care - no active intervention
- Combination Treadmill training group (Experimental): Subjects randomized to Combination therapy received 20 minutes of Lokomat assisted treadmill training followed by up to 20 minutes of BWS treadmill training (without robotic assistance) twice a week.
  Interventions: Other: Body-weight supported treadmill training +/- Lokomat assistance

INTERVENTIONS:
Other: Body-weight supported treadmill training +/- Lokomat assistance — walking
  Other Names: Lokomat
  Arms: Combination Treadmill training group
Other: Usual Care - no active intervention — No treatment used for comparison
  Other Names: control group
  Arms: Control group

SUMMARY:
This study is being done to test the possible benefits of gait-specific training using body-weight supported, Lokomat assisted, treadmill training in people with Multiple Sclerosis.

ELIGIBILITY:
Main Inclusion Criteria:

* Clinical diagnosis of MS
* EDSS level between 3.5-6.0
* Problems with ambulation
* able to ambulate 25 feet without an assistive device

Main Exclusion Criteria:

* Lower extremity injuries that limit range of motion or function
* Unable to demonstrate an understanding of the process of the study and or fully understand instructions in order to safely participate in the study and use study equipment
* Body weight over 150 kg

  * complete inclusion/exclusion criteria listed in consent form

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2008-02; Primary Completion 2011-10 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Gait Parameters | Baseline, throughout study enrollment and 2 months follow-up

OTHER OUTCOMES:
6 minute walk | Baseline, throughout study enrollment and 2 months follow-up
  The 6 minute walk test is measured on a treadmill. The subject is asked to indicate the most comfortable treadmill speed to the therapist. The subject is instructed to walk as far as possible in 6 minutes and the total distance covered in 6 minutes is recorded. A harness, without body-weight support, is attached for safety.
MSQLI (Multiple Sclerosis Quality of Life Index) | Baseline, throughout study enrollment and 2 months follow-up
  The MSQLI is a battery consisting of 10 individual scales providing a quality of life measure that is both generic and MS-specific (Fischer et al, 1999). The MS quality of life index is a validated instrument used in accessing multiple aspects of quality of life for persons with MS. It is a modification of the short-form health survey (SF-36) and requires about 30-45 minutes to complete.
Timed 25-foot walk | Baseline, throughout study enrollment and 2 months follow-up
  Will be collected over-ground and on a straight 25-foot GaitRite electronic mat. The subject will be timed over the 25-foot distance both at their self-designated usual pace and at the fastest safe pace possible. Data will be collected using a laptop computer. The GaitRite system has software to calculate several measures including velocity, stride length, base width and number of steps.
Frequency of Falls | Baseline, throughout study enrollment and 2 months follow-up
  Falls will be recorded by the subjects onto a "Falls Calender" provided to the subjects. Subjects will be given the following definition of a fall: "an event which results in a person coming to rest inadvertently on the ground or other lower level, and other than as a consequence of the following: sustaining a violent blow; loss of consciousness; sudden onset of paralysis, as in a stroke and an epileptic seizure" (Vellas 1992).
FRT (Functional Reach Test) | Baseline, throughout study enrollment and 2 months follow-up
  The Functional Reach test is a measure of balance and is the difference from arm's length and maximal forward reach. The support case is fixed. The test utilizes a 48-inch measuring device or "yardstick" for measuring functional reach. Data is measured in inches (Duncan P. W. et al 1990).
CDP (Computerized Dynamic Posturography) | Baseline, throughout study enrollment and 2 months follow-up
  NeuroCom Smart Balance Master system. The use of CDP has allowed clinicians to objectively measure the postural components of balance (Liston 1996). CDP assesses sway by measuring shifts in the center of gravity (COG) as a person moves within the available limits of stability (LOS). Two types of tests will be used with CDP; they are the Sensory Organization Test (SOT) and the LOS test.
  1. SOT: measures sway and is designed to quantify an individual's ability to maintain balance in a variety of complex sensory conditions.
  2. LOS: measures volitional control of the COG. Test measures include maximum end-point excursion for anterior, posterior, right, and left movements.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Lo, MD, PhD, Principal Investigator — Mandell Center for Multiple Sclerosis at Mount Sinai Rehabilitation Hospital
Locations (1):
- Mandell Center for Multiple Sclerosis at Mt. Sinai Rehabilitation Hospital, Hartford, Connecticut, United States

REFERENCES:
- [Background] Fischer JS, LaRocca NG, Miller DM, Ritvo PG, Andrews H, Paty D. Recent developments in the assessment of quality of life in multiple sclerosis (MS). Mult Scler. 1999 Aug;5(4):251-9. doi: 10.1177/135245859900500410. PMID 10467384
- [Background] Vellas B, Baumgartner RN, Wayne SJ, Conceicao J, Lafont C, Albarede JL, Garry PJ. Relationship between malnutrition and falls in the elderly. Nutrition. 1992 Mar-Apr;8(2):105-8. PMID 1591453
- [Background] Duncan PW, Weiner DK, Chandler J, Studenski S. Functional reach: a new clinical measure of balance. J Gerontol. 1990 Nov;45(6):M192-7. doi: 10.1093/geronj/45.6.m192. PMID 2229941
- [Background] Liston RA, Brouwer BJ. Reliability and validity of measures obtained from stroke patients using the Balance Master. Arch Phys Med Rehabil. 1996 May;77(5):425-30. doi: 10.1016/s0003-9993(96)90028-3. PMID 8629916
- See also: Mandell Center for Multiple Sclerosis home page — http://www.saintfrancisdoctors.com/ms